CLINICAL TRIAL: NCT05442060
Title: A Randomized, Open-Label, Phase 2 Study to Evaluate OBI-833/OBI-821 in Combination With First-Line Erlotinib in Patients With EGFR-Mutated, Globo H-Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: To Evaluate OBI-833/OBI-821 in Combination With First-Line Erlotinib in Patients With EGFR-Mutated, Globo H-Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: EGFR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OBI-833-003
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: OBI-833/OBI-821; Erlotinib; EGFR-Mutated; Globo H; Globo H positive; Locally advanced non-small cell lung cancer; Metastatic non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erlotinib (Active Comparator): Erlotinib (150 mg daily)
  Interventions: Drug: Erlotinib (150 mg daily)
- Erlotinib + OBI-833/OBI-821 (Experimental): Erlotinib (150 mg daily) + 30 μg OBI-833/100 μg OBI-821
  Interventions: Biological: 30 μg OBI-833/100 μg OBI-821; Drug: Erlotinib (150 mg daily)

INTERVENTIONS:
Biological: 30 μg OBI-833/100 μg OBI-821 — Each subject in the OBI-833/OBI-821 + erlotinib combination arm will be treated with OBI-833/OBI-821 weekly for 4 doses (Weeks 1, 2, 3, 4), then every 2 weeks for 2 doses (Weeks 6, 8), then every 4 weeks for 4 doses (Weeks 12, 16, 20, 24), and then every 8 weeks until documented disease progression, intolerable adverse events (AEs)/toxicity, consent withdrawal, death, loss to follow-up, or up to 80 weeks from randomization.
  Arms: Erlotinib + OBI-833/OBI-821
Drug: Erlotinib (150 mg daily) — All subjects in both arms will continue to receive erlotinib as the background therapy (150 mg daily).

SUMMARY:
This study is a randomized, active control, open-label, phase 2 trial. Erlotinib-treated NSCLC patients will be screened for Globo H, and only Globo H+ (H score ≥ 100) subjects are eligible for the study. Eligible subjects who have been treated with 3±1 months of first-line erlotinib and have achieved stable disease (SD) or partial response (PR) status will be randomized in the ratio of 1:1 to receive erlotinib alone or erlotinib plus OBI-833/OBI-821 therapy.

DETAILED DESCRIPTION:
All subjects in both arms will continue to receive erlotinib as the background therapy. Each subject in the OBI-833/OBI-821 + erlotinib combination arm will be treated with OBI-833/OBI-821 weekly for 4 doses (Weeks 1, 2, 3, 4), then every 2 weeks for 2 doses (Weeks 6, 8), then every 4 weeks for 4 doses (Weeks 12, 16, 20, 24), and then every 8 weeks until documented disease progression, intolerable adverse events (AEs)/toxicity, consent withdrawal, death, loss to follow-up, or up to 80 weeks from randomization. Subjects in the OBI-833/OBI-821 + erlotinib arm will be evaluated for humoral immune responses until disease progression. Upon completion of or discontinuation from the study treatment, all subjects will be followed up for survival by phone call every 3 months until up to 12 months after the end of treatment (EoT) visit.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 20 years.
2. Pathologically or cytologically confirmed diagnosis of non-small cell lung cancer whose stage is IIIB, IIIC, IVA, or IVB according to the AJCC Cancer Staging System, 8th Edition.
3. The tumor harbors an exon 19 deletion or exon 21 L858R mutation in EGFR, confirmed locally.
4. Patient must have a documented Globo H H-score of at least 100 using a validated central IHC assay.
5. Patient must have received 3±1 months of first-line erlotinib therapy under a stable dosage of 150 mg/day, have achieved SD or PR before randomization (as confirmed by the Investigator), and plan to continue the erlotinib treatment at 150 mg/day.
6. At least one measurable tumor lesion according to RECIST version 1.1 as assessed by the Investigator (local radiological image assessment).
7. Life expectancy ≥ 6 months.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Organ Function Requirements - Subjects must have adequate organ functions as defined below:

   * AST/ALT ≤ 3X ULN (upper limit of normal); AST/ALT ≤ 5X ULN in the presence of liver metastases
   * Total bilirubin ≤ 2.0 X ULN
   * Serum creatinine ≤ 1.5X ULN
   * ANC ≥ 1,500 /µL
   * Platelets ≥ 100,000/µL
10. All eligible patients of childbearing potential must use effective contraception during study treatment, and for at least 2 months after the last dose of OBI-833/OBI-821 and for at least 2 weeks after the last dose of erlotinib. Subjects not of childbearing potential (i.e., permanently sterilized, postmenopausal) can be included in the study. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.
11. Understand and provide a written informed consent document according to institutional guidelines.

Exclusion Criteria:

1. Patient who has CNS metastasis.
2. Patient who is pregnant or breast-feeding at entry.
3. Patient with splenectomy.
4. Patient with HIV infection, active hepatitis B infection, or active hepatitis C infection.
5. Patient with a positive test result for SARS-CoV-2 detected by standard reverse transcription-polymerase chain reaction (RT-PCR) at screening.
6. Patient with any autoimmune or other disorders requiring IV/oral steroids or immunosuppressive or immunomodulatory therapies.

   (e.g., type 1 juvenile onset diabetes mellitus, antibody positive for rheumatoid arthritis, Graves disease, Hashimoto thyroiditis, lupus, scleroderma, systemic vasculitis, hemolytic anemia, immune mediated thrombocytopenia, Crohn disease, ulcerative colitis, and psoriasis).
7. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Grade 0 or 1 (using National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0), except for alopecia and laboratory values listed in the inclusion criteria.
8. A history of other malignancies (except non-melanoma skin carcinoma, carcinoma in situ of the uterine cervix, follicular or papillary thyroid cancer) within 5 years prior to randomization.
9. Patient with any known uncontrolled comorbid illness including ongoing or active infections, symptomatic congestive heart failure (NYHA>2), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Treatment with any of the following therapies within 4 weeks prior to randomization:

    * Anti-cancer therapies, including chemotherapy and targeted therapy (except erlotinib).
    * Radiotherapy.
    * Immunotherapy, including monoclonal antibodies, cytokines, interferons, and checkpoint inhibitors.
    * Immunosuppressants, including cyclosporin, rapamycin, tacrolimus, rituximab, alemtuzumab, natalizumab, and cyclophosphamide.
    * Other biologics, including G-CSF and other hematopoietic growth factors.
    * Live attenuated vaccines.
    * IV/oral steroids except single prophylactic use in CT/MRI scan or other one-time use in approved indications. Use of inhaled and topical (except on the injection site) steroids is allowed.
    * Alternative and complementary medicine that may affect the immune system.
    * Other investigational drugs.
11. Subject with pleural effusions and/or ascites, due to malignancy, requiring paracentesis every 2 weeks or more frequently.
12. Subject with any known severe allergies (e.g., anaphylaxis) to any active or inactive ingredients in the study drugs.
13. Any other reason that the investigator deems the patient to be unsuitable for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rated at one year | One year
  One year progression-free survival rated by RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Lance Ou, Study Director — OBI Pharma, Inc
Locations (7):
- Taiwan (7):
  - Taipei Veterans General Hospital, Taipei, Beitou District
  - National Taiwan University Cancer Center, Taipei, Da'an Dist.
  - Linkou Chang Gung Memorial Hospital, Taoyuan District, Guishan Dist.
  - Tri-Service General Hospital, Taipei, Neihu District
  - Shuang Ho Hospital, New Taipei City, Zhonghe District
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist.
  - Taichung Veterans General Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No